CLINICAL TRIAL: NCT05736861
Title: ACTIV-6: COVID-19 Outpatient Randomized Trial to Evaluate Efficacy of Repurposed Medications
Brief Title: ACTIV-6: COVID-19 Study of Repurposed Medications - Arm A (Ivermectin 400)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Susanna Naggie, MD (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Susanna Naggie, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00107921_A; 3U24TR001608-05W1 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-02-21 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID-19; ivermectin; Placebo; Duke University Health System; Outcomes; Duke Clinical Research Institute; ACTIV 6; ACTIV
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled, Randomized Trial
Who Masked: Participant, Care Provider
Masking Description: The participant and study teams will know which study drug the participant is allocated to, but will be blinded to study drug versus placebo because they will be matching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Ivermectin 400 (Experimental): Ivermectin - 7-mg tablets
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight for a daily dose of approximately 300-400 µg/kg.
  Interventions: Drug: Ivermectin
- Arm A - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight, matched to active study drug dosing.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — Each participant will receive a sufficient quantity of 7-mg tablets to be taken as directed based on their weight. The tablets are white, round, biconvex tablets with "123" over the scoring on one side. All packaging will be labeled to indicate that the product is for investigational use.
  Other Names: Ivermectin Tablets
  Arms: Arm A - Ivermectin 400
Other: Placebo — Each study arm will contain a placebo comparator. Placebo will look similar to study drug and will be administered via the same route of administration and dose. However, placebo will be an inactive substance, containing no study drug.
  Arms: Arm A - Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of repurposed medications (study drug(s) in reducing symptoms of non-hospitalized participants with mild to moderate COVID-19. Participants will receive either study drug or placebo. They will self-report any new or worsening symptoms or medical events they may experience while taking study drug or placebo. This study is intended to be all remote with no in person visits, unless the study team feels it is in the best interest of a participant to see them in person.

Prior and current drug arms are listed on clinicaltrials.gov and will be updated with the activation of any new drug arms. This protocol was originally registered under NCT04885530. Per recent guidance on reporting master protocol research programs (MPRPs), a separate record for Arm A was created.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel betacoronavirus that first emerged in December 2019 and has since caused a global pandemic unseen in almost a century with respect to the number of cases and overall mortality. The clinical disease related to SARS-CoV-2 is referred to as Coronavirus Disease 2019 (COVID-19). Over 2020, advances were made for treatment of COVID-19 and several vaccinations have received emergency use authorization for prevention of SARS-CoV-2 infections. However, the pandemic continues to evolve with new variants and surges of infections in different regions of the world, requiring an ongoing evidence-generating platform, in particular for the treatment of COVID-19 infection in the outpatient setting.

This proposed platform protocol can serve as an evidence generating system for prioritized drugs repurposed from other indications with an established safety record and preliminary evidence of clinical efficacy for the treatment of COVID-19. The ultimate goal is to evaluate if repurposed medications can make participants feel better faster and reduce death and hospitalization.

This platform protocol is designed to be flexible so that it is suitable for a wide range of settings within healthcare systems and in community settings where it can be integrated into routine COVID-19 testing programs and subsequent treatment plans. This platform protocol will enroll participants in an outpatient setting with a confirmed polymerase chain reaction (PCR) or antigen test for SARS-CoV-2.

Participants will be randomized to study drugs or placebo based on the arms that are actively enrolling at the time of randomization. Study drugs may be added or removed according to adaptive design and/or emerging evidence. When there are multiple study drugs available, randomization will occur based on appropriateness of each drug for the participant as determined by the study protocol and investigator and participant equipoise. Each participant will be required to randomize to at least one study drug versus placebo. The probability of placebo to treatment will remain the same regardless of eligibility decisions.

Eligible participants will be randomized (1:1), in a blinded fashion, to either the study drug arm or placebo arm in addition to standard of care. As additional study drugs are added, the randomization will be altered to leverage placebo data across arms. Participants will receive a complete supply study drug or placebo with the quantity depending on the study drug/placebo to which they are randomized.

All study visits are designed to be remote. However, screening and enrollment may occur in-person at sites and unplanned study visits may occur in-person or remotely, as deemed appropriate by the site investigator for safety purposes. Participants will be asked to complete questionnaires and report safety events during the study. Participants will be prompted by the online system to report safety events and these will be reviewed and confirmed via medical records and site staff, as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Completed Informed Consent
* Age ≥ 30 years old
* Confirmed SARS-CoV-2 infection by any authorized or approved polymerase chain reaction (PCR) or antigen test collected within 10 days of screening
* Two or more current symptoms of acute infection for ≤7 days. Symptoms include the following: fatigue, dyspnea, fever, cough, nausea, vomiting, diarrhea, body aches, chills, headache, sore throat, nasal symptoms, new loss of sense of taste or smell

Exclusion Criteria:

* Prior diagnosis of COVID-19 infection (> 10 days from screening)
* Current or recent (within 10 days of screening) hospitalization
* Current use of study drug or study drug/device combination*
* Known allergy/sensitivity or any hypersensitivity to components of the study drug or placebo*
* Known contraindication(s) to study drug including prohibited concomitant medications*

[If only one study drug appendix is open at the time of enrollment. If multiple study drug appendices are open, a participant may opt-out of any study drug appendix or be excluded from any study drug appendix based on contraindications listed in the study drug appendix, current use of study drug, or known allergy/sensitivity/hypersensitivity and still remain eligible for the remaining study drug appendices.]

Arm-specific exclusion criteria:

* End-stage renal disease on renal replacement therapy
* Liver failure or decompensated cirrhosis
* Use of warfarin, CYP3A4, P-gp inhibitor drugs, or CYP3A4 substrates
* Nursing mothers
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Naggie, MD, Principal Investigator — Duke Clinical Research Institute; Adrian Hernandez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (87):
- United States (87):
  - Lamb Health, LLC, Gilbert, Arizona
  - First Care Medical Clinic, Mesa, Arizona
  - Trident Health Center, Peoria, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Assuta Family Medical Group APMC, North Hollywood, California
  - Stanford, Palo Alto, California
  - Doctors Medical Group of Colorado Springs, P.C., Colorado Springs, Colorado
  - Pine Ridge Family Medicine Inc., Colorado Springs, Colorado
  - Tabitha B. Fortt, M.D., LLC, Stamford, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Lupus Foundation of Gainesville, Gainesville, Florida
  - University of Florida Health, Gainesville, Florida
  - University of Florida-JAX-ASCENT, Jacksonville, Florida
  - AMRON Vitality and Wellness Center, LLC, Jacksonville, Florida
  - Sunshine Walk In Clinic, Lake Mary, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Innovation Clinical Trials Inc., Palmetto Bay, Florida
  - Lice Source Services Plantation, Plantation, Florida
  - Premier Health, St. Petersburg, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - UF Health Precision Health Research, The Villages, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Essential Medical Care, Inc., College Park, Georgia
  - David Kavtaradze MD, Inc., Cordele, Georgia
  - Elite Family Practice, Douglasville, Georgia
  - Christ the King Health Care, P.C., Loganville, Georgia
  - Miller Family Practice, LLC, Macon, Georgia
  - Olivo Wellness Medical Center, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Advanced Medical Care, Ltd, Lake Zurich, Illinois
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Del Pilar Medical and Urgent Care, Mishawaka, Indiana
  - University of Kansas - Wichita, Wichita, Kansas
  - A New Start II, LLC, Central City, Kentucky
  - University Medical Center- New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Rockville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Health Quality Primary Care, Lawrence, Massachusetts
  - Ananda Medical Clinic, Dearborn, Michigan
  - GFC of Southeastern Michigan, PC, Detroit, Michigan
  - Romancare Health Services, Detroit, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri - Columbia, Columbia, Missouri
  - Comprehensive Pain Management and Endocrinology, Henderson, Nevada
  - Focus Clinical Research Solutions, Bayonne, New Jersey
  - Raritan Bay Primary Care & Cardiology Associates, Matawan, New Jersey
  - Mediversity Healthcare, Turnersville, New Jersey
  - Geriatrics and Medical Associates, Clinton, New York
  - Weill Cornell Medical College, New York, New York
  - Spinal Pain and Medical Rehab, PC, Yonkers, New York
  - Vaidya MD PLLC, Clayton, North Carolina
  - Maria Medical Center, PLLC, Dunn, North Carolina
  - Duke Clinical Research Institute, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Diabetes and Endocrinology Assoc. of Stark County, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - TriHealth, Inc, Montgomery, Ohio
  - The Heart and Medical Center, Durant, Oklahoma
  - Hugo Medical clinic, Hugo, Oklahoma
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Trials Center of Middle TN, Franklin, Tennessee
  - Rapha Family Wellness, Hendersonville, Tennessee
  - Medical Specialists of Knoxville, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Express Family Clinic, Allen, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - Highlands Medical Associates, P.A., Highlands, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Family Practice Doctors P.A., Humble, Texas
  - Vytalus Medical Group, Humble, Texas
  - Texas Health Physicians Group, Irving, Texas
  - University Diagnostics and Treatment Clinic, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Jeremy W. Szeto, D.O., P.A., Sugar Land, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
We will share this data after it has been de-identified. We will share data beginning around 6 months after publication and for up to 36 months afterward. Access will only be shared with those who have obtained prior IRB approval to be able to access this data.
Supporting Information: SAP, CSR
Time Frame: Up to 36 months after publication
Access Criteria: Interested investigators will need to seek prior IRB approval before access to any data is granted.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Ivermectin 400: Ivermectin - 7-mg tablets
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight for a daily dose of approximately 300-400 µg/kg.
  Ivermectin: Each participant will receive a sufficient quantity of 7-mg tablets to be taken as directed based on their weight. The tablets are white, round, biconvex tablets with "123" over the scoring on one side. All packaging will be labeled to indicate that the product is for investigational use.
- Arm A - Placebo: Placebo - appearance and size matched to active study drug.
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight, matched to active study drug dosing.
  Placebo: Each study arm will contain a placebo comparator. Placebo will look similar to study drug and will be administered via the same route of administration and dose. However, placebo will be an inactive substance, containing no study drug.
Period: Overall Study
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Started | 919 | 881
Completed | 817 | 774
Not Completed | 102 | 107

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo | Total
Number analyzed (Participants) | 817 | 774 | 1591
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [39 to 56] | 48 [39 to 56] | 47 [39 to 56]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 508 | 424 | 932
  Sex/Gender: Male | 309 | 349 | 658
  Sex/Gender: Prefer Not to Answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 70 | 163
  Not Hispanic or Latino | 724 | 704 | 1428
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 5 | 16
  Asian | 14 | 16 | 30
  Black, African American, or African | 50 | 53 | 103
  Middle Eastern or North African | 29 | 23 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  White | 643 | 619 | 1262
  More than one race | 19 | 8 | 27
  None of the above | 25 | 16 | 41
  Prefer not to answer | 14 | 24 | 38
  No response | 12 | 7 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 817 | 774 | 1591

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Recovery in Days
Description: Time to sustained recovery was the number of days between receipt of study drug and the third of 3 consecutive days without symptoms. Participants who died, by definition, did not recover regardless of reported symptom freedom. The reported summary is the median survival time.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
days | 12 [11 to 13] | 13 [12 to 14]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority — Decision rule based on Bayesian posterior probability of efficacy. The decision threshold was a posterior probability of 0.95. A prespecified skeptical prior for the treatment effect was used to preserve type I error below 0.05; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.96 to 1.17] — The interval is a highest-density credible interval. Adjustment variables: randomization, age, sex, duration of symptoms prior to study drug, calendar time, vaccination status, geographic region, call center indicator, and baseline symptom severity

2. Secondary Outcome: Number of Participants With Hospitalization or Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
Participants | 10 | 9
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.4 to 2.6] — The interval is a highest-density credible interval. Descriptive analysis is a maximum partial likelihood proportional hazards regression model. Low event rate precluded covariate adjustment

3. Secondary Outcome: Number of Participants With Mortality
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
Participants | 1 | 0

4. Secondary Outcome: Time to Mortality
Description: Time to mortality was the number of days between drug receipt and death.
Time Frame: Up to 28 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
days | NA [NA to NA] — Per the protocol/SAP, this endpoint is only analyzed if the number of total events exceeds 30. Due to the low event rate, the statistical analysis was not completed. | NA [NA to NA] — Per the protocol/SAP, this endpoint is only analyzed if the number of total events exceeds 30. Due to the low event rate, the statistical analysis was not completed.

5. Secondary Outcome: Number of Participants With Hospitalization, Urgent Care, Emergency Room Visit, or Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
Participants | 32 | 28
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority — Statistical analysis was a Bayesian proportional hazards regression model with covariate adjustment and weakly informative priors; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.6 to 1.8] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 7
Description: COVID Clinical Progression Scale is a scale of 0 to 8 where 0 = No clinical or virological evidence of infection, 1 = No limitation of activities, 2 = Limitation of activities, 3 = Hospitalized, no oxygen therapy, 4 = Hospitalized, on oxygen by mask or nasal prongs, 5 = Hospitalized, on non-invasive ventilation or high-flow oxygen, 6 = Hospitalized, on intubation and mechanical ventilation, 7 = Hospitalized, on ventilation + additional organ support (pressors, RRT, ECMO), 8 = Death.
Time Frame: Day 7
Population: Data not collected on 9 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 813 | 769
Participants
  0 = No clinical or virological evidence of infection | 45 | 51
  1 = No limitation of activities | 708 | 646
  2 = Limitation of activities | 53 | 68
  3 = Hospitalized, no oxygen therapy | 0 | 1
  4 = Hospitalized, on oxygen by mask or nasal prongs | 5 | 2
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 0 | 1
  6 = Hospitalized, on intubation and mechanical ventilation | 1 | 0
  7 = Hospitalized, on ventilation + additional organ support (pressors, RRT, ECMO) | 0 | 0
  8 = Death | 1 | 0
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority — Statistical analysis was a Bayesian cumulative probability ordinal regression model with covariate adjustment and weakly informative priors; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.50 to 1.13] — The interval is a highest-density credible interval on the log relative odds scale. Odds ratio estimate from a Bayesian cumulative probability ordinal regression model with weakly informative priors

7. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 14
Description: as for outcome 6
Time Frame: Day 14
Population: Data not collected on 21 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 805 | 765
Participants
  0 = No clinical or virological evidence of infection | 52 | 60
  1 = No limitation of activities | 722 | 664
  2 = Limitation of activities | 28 | 38
  3 = Hospitalized, no oxygen therapy | 0 | 1
  4 = Hospitalized, on oxygen by mask or nasal prongs | 0 | 1
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 1 | 1
  6 = Hospitalized, on intubation and mechanical ventilation | 1 | 0
  7 = Hospitalized, on ventilation + additional organ support (pressors, RRT, ECMO) | 0 | 0
  8 = Death | 1 | 0
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.39 to 1.13] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Number of Participants at Each Score on the COVID Clinical Progression Scale at Day 28
Description: as for outcome 6
Time Frame: Day 28
Population: Data not collected on 36 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 795 | 760
Participants
  0 = No clinical or virological evidence of infection | 56 | 59
  1 = No limitation of activities | 718 | 682
  2 = Limitation of activities | 19 | 18
  3 = Hospitalized, no oxygen therapy | 0 | 1
  4 = Hospitalized, on oxygen by mask or nasal prongs | 0 | 0
  5 = Hospitalized, on non-invasive ventilation or high-flow oxygen | 0 | 0
  6 = Hospitalized, on intubation and mechanical ventilation | 1 | 0
  7 = Hospitalized, on ventilation + additional organ support (pressors, RRT, ECMO) | 0 | 0
  8 = Death | 1 | 0
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.52 to 1.91]; The interval is a highest-density credible interval on the log relative odds scale. Odds ratio estimate from a Bayesian cumulative probability ordinal regression model with weakly informative priors

9. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Physical Function
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a higher score correlates to better outcome for physical function.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 763 | 715
  Day 7 | 19 [16 to 20] | 19 [16 to 20]
  Day 14: number analyzed (Participants) | 753 | 707
  Day 14 | 20 [18 to 20] | 20 [18 to 20]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 20 [20 to 20] | 20 [20 to 20]
  Day 90: number analyzed (Participants) | 714 | 685
  Day 90 | 20 [20 to 20] | 20 [20 to 20]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.82 to 1.25] — Initially estimated on the log relative odds scale, and then transformed to the odds ratio scale. On the log relative odds scale, the estimated parameter value was the posterior mean. Interval estimate is symmetric density Bayesian credible interval
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.78 to 1.23] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.82 to 1.41] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.57 to 1.01] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Fatigue
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for fatigue.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 715
  Day 7 | 9 [7 to 13] | 9 [7 to 13]
  Day 14: number analyzed (Participants) | 752 | 707
  Day 14 | 7 [4 to 9] | 7 [4 to 9]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 5 [4 to 8] | 5 [4 to 8]
  Day 90: number analyzed (Participants) | 714 | 685
  Day 90 | 4 [4 to 8] | 4 [4 to 8]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.92 to 1.32] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.83 to 1.22] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.83 to 1.24] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.72 to 1.10]; Initially estimated on the log relative odds scale, and then transformed to the odds ratio scale. On the log relative odds scale, the estimated parameter value was the posterior mean. Interval estimate is symmetric density Bayesian credible interval

11. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Pain
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for pain.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 715
  Day 7 | 5 [4 to 9] | 5 [4 to 8]
  Day 14: number analyzed (Participants) | 751 | 706
  Day 14 | 4 [4 to 7] | 4 [4 to 7]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 4 [4 to 5] | 4 [4 to 4]
  Day 90: number analyzed (Participants) | 714 | 685
  Day 90 | 4 [4 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.80 to 1.20] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.78 to 1.25] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.86 to 1.43] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.66 to 1.12] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Depression
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20, where a lower score correlates to better outcome for depression.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 715
  Day 7 | 4 [4 to 6] | 4 [4 to 6]
  Day 14: number analyzed (Participants) | 752 | 706
  Day 14 | 4 [4 to 5] | 4 [4 to 5]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 4 [4 to 5] | 4 [4 to 5]
  Day 90: number analyzed (Participants) | 713 | 685
  Day 90 | 4 [4 to 5] | 4 [4 to 5]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.87 to 1.35] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.96 to 1.57] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.92 to 1.54] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.71 to 1.18] — [estimate comment as in outcome 9, analysis 1]

13. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Anxiety
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a lower score correlates to better outcome for anxiety.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 714
  Day 7 | 5 [4 to 8] | 5 [4 to 8]
  Day 14: number analyzed (Participants) | 752 | 706
  Day 14 | 4 [4 to 6] | 4 [4 to 6]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 4 [4 to 6] | 4 [4 to 5]
  Day 90: number analyzed (Participants) | 713 | 685
  Day 90 | 4 [4 to 5] | 4 [4 to 5]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.97 to 1.47] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.84 to 1.33] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.95 to 1.55] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.73 to 1.19] — [estimate comment as in outcome 9, analysis 1]

14. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Social
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a higher score correlates to better outcome for social roles and activities.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 715
  Day 7 | 17 [13 to 20] | 17 [13 to 20]
  Day 14: number analyzed (Participants) | 752 | 705
  Day 14 | 20 [16 to 20] | 20 [16 to 20]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 20 [17 to 20] | 20 [17 to 20]
  Day 90: number analyzed (Participants) | 714 | 684
  Day 90 | 20 [17.25 to 20] | 20 [18 to 20]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.86 to 1.26] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.85 to 1.29] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.85 to 1.34] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.80 to 1.28] — [estimate comment as in outcome 9, analysis 1]

15. Secondary Outcome: Quality of Life (QOL) as Measured by the PROMIS-29 - Sleep Domain
Description: The PROMIS-29 (Patient-Reported Outcomes Measurement Information System) consists of seven health domains with four 5-level items associated with each and a pain intensity assessment using a 0-10 numeric rank. The seven health domains include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. Raw score ranges from 4-20 where a lower score correlates to better outcome for sleep.
Time Frame: Day 7, 14, 28, and 90
Population: Participants who responded to the quality of life survey at each timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
score on a scale
  Day 7: number analyzed (Participants) | 764 | 715
  Day 7 | 10 [8 to 12] | 10 [7 to 12]
  Day 14: number analyzed (Participants) | 752 | 705
  Day 14 | 9 [6 to 12] | 9 [6 to 11]
  Day 28: number analyzed (Participants) | 742 | 704
  Day 28 | 8 [6 to 11] | 9 [6 to 11]
  Day 90: number analyzed (Participants) | 714 | 685
  Day 90 | 8 [6 to 11] | 8 [6 to 11]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 7; Test type: Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.88 to 1.27] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 14; Test type: Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.79 to 1.14] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 28; Test type: Other; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.75 to 1.09] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Day 90; Test type: Other; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.93 to 1.36] — [estimate comment as in outcome 9, analysis 1]

16. Secondary Outcome: Time Unwell in Days as Measured by the Symptom and Clinical Event Scale
Description: The symptom and clinical event scale is a daily measurement that combines the global symptom burden scale with clinical events hospitalization and mortality. (No symptoms, mild symptoms, moderate symptoms, severe symptoms, hospitalized, deceased). Time unwell was the portion of follow-up (in days) that a participant was symptomatic, hospitalized, or deceased. The quantity is estimated from a Bayesian longitudinal ordinal regression model with covariate adjustment and weakly informative priors.
Time Frame: Up to 14 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
days | 10.96 [10.78 to 11.15] | 11.45 [11.28 to 11.60]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Test type: Superiority; Difference in model estimate time unwell = -0.49, 95% CI 2-sided [-0.82 to -0.15] — The interval is a highest-density credible interval

17. Secondary Outcome: Mean Days Benefit as Measured by the Symptom and Clinical Event Scale
Description: The symptom and clinical event scale is a daily measurement that combines the global symptom burden scale with clinical events hospitalization and mortality. (No symptoms, mild symptoms, moderate symptoms, severe symptoms, hospitalized, deceased). The cumulative benefit of treatment A is the probability of experiencing a better outcome on treatment A compared to treatment B, summed over the days of follow-up. The difference between the cumulative benefit of treatment A and the cumulative benefit of treatment B is known as the difference in days benefit. Measure of dispersion is 95% credible interval.
Time Frame: Up to 14 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
Number analyzed (Participants) | 817 | 774
days | 3.91 [3.69 to 4.13] | 3.31 [3.11 to 3.51]
Statistical Analysis 1: Comparison: Arm A - Ivermectin 400 vs Arm A - Placebo; Analysis is exploratory. No hypothesis test or decision rule was evaluated; Test type: Superiority; Difference in model estimated means = 0.59, 95% CI 2-sided [0.18 to 0.99] — The interval is a highest-density credible interval

ADVERSE EVENTS:
Time Frame: Up to 90 days
Description: Participants were asked to complete daily assessments and report adverse events via the study portal through day 14, then at other intervals through day 28, and at the final study visit at day 90.
  Adverse event tables were updated on 5/16/2023 to reflect data cleaning and data monitoring efforts by contributing sites. Some sites determined that some previously reported events should not have been reported per the criteria noted in the protocol.
Arm/Group | Arm A - Ivermectin 400 | Arm A - Placebo
All-Cause Mortality (participants affected / at risk) | 1/817 | 0/774
Serious Adverse Events (participants affected / at risk) | 13/817 | 17/774
Other Adverse Events (participants affected / at risk) | 16/817 | 13/774
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Ivermectin 400 (N=817) | Arm A - Placebo (N=774)
COVID-19 pneumonia (Infections and infestations) | 3 | 4
COVID-19 pneumonia aggravated (Infections and infestations) | 0 | 3
Bacteremia, with signs and symptoms (Infections and infestations) | 0 | 1
Pneumonia due to Staphylococcus (Infections and infestations) | 1 | 0
Pneumonia due to Streptococcus, group b (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Viral bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Venous thromboembolism (Vascular disorders) | 0 | 2
Diplopia (Eye disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute Cholecystitis (Hepatobiliary disorders) | 1 | 0
Coronary vasospasm (Vascular disorders) | 0 | 1
COVID-19 pneumonia worsening (Infections and infestations) | 1 | 0
Death due to COVID-19 (Infections and infestations) | 1 | 0
Opthalmic migraine (Eye disorders) | 0 | 1
Pneumonia due to COVID-19 virus (Infections and infestations) | 1 | 0
Upper GI bleed (Vascular disorders) | 0 | 1
Worsening of covid-19 pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Ivermectin 400 (N=817) | Arm A - Placebo (N=774)
Accelerated hair loss (Skin and subcutaneous tissue disorders) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1
Blood pressure raised (Investigations) | 1 | 0
Chest tightness (General disorders) | 0 | 1
Confusion (Nervous system disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dyspnea (Cardiac disorders) | 1 | 0
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0
Hepatic steatosis (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Insomnia (Nervous system disorders) | 0 | 1
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Nausea and emesis (Gastrointestinal disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seasonal Allergies (Immune system disorders) | 0 | 1
Shoulder dislocation (Injury, poisoning and procedural complications) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus infection (Infections and infestations) | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Suspected Covid-19 (Infections and infestations) | 0 | 1
Tiredness (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT05736861/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05736861/ICF_001.pdf